CLINICAL TRIAL: NCT05100849
Title: Efficacy of Kinect-based Versus Tablet-based Cognitive Training Through Simulations of Instrumental Activities of Daily Living: a Pilot Study With Chronic Psychiatric Patients
Brief Title: Kinect-based Versus Tablet-based Cognitive Training: a Pilot Study With Psychiatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Collaborators: Casa de Saúde Câmara Pestana (Unknown)
Responsible Party: Principal Investigator, Sergi Bermúdez i Badia, Associate Professor at the University of Madeira and Senior Researcher at NOVA LINCS, Universidade da Madeira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/2021
Record Dates: First submitted 2021-05-27; First posted 2021-10-29 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Psychiatric Disorder
Keywords: Cognitive training; Simulations of instrumental activities of daily living; Tablet-based cognitive training; Kinect-based cognitive training; Psychiatric disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinect-based cognitive training (Experimental): Standard treatment protocol and 14 sessions (biweekly during 30 minutes) of Kinect-based cognitive training inspired by instrumental activities of daily living.
  Interventions: Procedure: Kinect-based cognitive training
- Tablet-based cognitive training (Experimental): Standard treatment protocol and 14 sessions (biweekly during 30 minutes) of Tablet-based cognitive training inspired by instrumental activities of daily living.
  Interventions: Procedure: Tablet-based cognitive training

INTERVENTIONS:
Procedure: Kinect-based cognitive training — The Kinect-based group will be involved in the standard treatment protocol and will perform a 14-sessions cognitive training program that consists of instrumental activities of daily living simulations. The cognitive training content will be projected onto a wall and patients will interact with the content, i.e., the selection of the appropriate response, through movement (kinect).
  Arms: Kinect-based cognitive training
Procedure: Tablet-based cognitive training — The Tablet-based group will be involved in the standard treatment protocol and will perform a 14-sessions cognitive training program that consists of instrumental activities of daily living simulations. Patients will interact with the cognitive training content through a tablet.
  Arms: Tablet-based cognitive training

SUMMARY:
This study aims to analyze which cognitive training experimental condition - Tablet versus Kinect - results in greater cognitive, mood, quality of life, and functional gains in a sample of chronic psychiatric patients.

DETAILED DESCRIPTION:
Cognitive deficits are a nuclear feature of several psychiatric disorders, leading to a decrease in functional abilities and quality of life. Besides facilitating the inclusion of more ecologically valid stimuli and training tasks, technology-based cognitive training methods allow more dynamic interactions with the cognitive training content, which can result in an enhancement of patients' motivation and engagement in the therapeutic process. The modality of interaction with the cognitive training content may influence patients' response to cognitive training interventions. For instance, cognitive training through the tablet requires essentially hand movements (e.g., interaction with the training tasks by touching the correct stimuli), while cognitive training through the Kinect involves the performance of wide range movements (e.g., interaction with the training tasks by making specific "body" movements to select the correct stimuli). This study aims to analyze which cognitive training experimental condition - Tablet versus Kinect - results in greater cognitive, mood, quality of life, and functional gains in a sample of chronic psychiatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric diagnosis;
* Maximum age: 75 years old;
* Relatively preserved language abilities (expressive and receptive language);
* Being able to read and write;
* Having no motor limitations;
* Having no medical history of neurological conditions (e.g., stroke, traumatic brain injury, multiple sclerosis, etc.)
* Preserved visual and auditory acuity;

Exclusion Criteria:

* Experiencing an acute psychiatric episode.

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) (Cognitive screening) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the Montreal Cognitive Assessment (MoCA); Min score=0; Max score=30; Higher scores mean a better outcome
Frontal Assessment Battery (FAB) (Executive functions screening) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the Frontal Assessment Battery (FAB). Min score=0; Max score=18; Higher scores mean a better outcome.
Toulouse-Piéron Cancellation Test (TP) (Sustained and selective attention) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the Toulouse-Piéron Cancellation Test (TP); Min score=0; Max score=dependent on patients' performance during a 10-min time frame; A higher work efficiency index means a better outcome, whereas a higher dispersion index means a worse outcome.
Rey Complex Figure Test (RCFT) (Visuospatial skills and visual memory) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the Rey Complex Figure Test (RCFT); Min score=0; Max score=36; Higher scores mean a better outcome.
Symbol Search and Coding (WAIS-III) (Processing speed) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the Symbol Search and Coding (WAIS-III); Min score=0; Max score dependent on patients' performance in a 120 seconds time frame. Higher scores in both subtests mean a better outcome.
Verbal Fluency Tests (semantic and phonemic) (Executive Functions) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the Verbal Fluency Tests (semantic and phonemic); Min score=0; Max score dependent on patients' performance during a 1-minute time frame. Higher scores on both verbal fluency tests mean a better outcome.
Free and Cued Selective Reminding Test (FCSRT) (Verbal Memory) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the Free and Cued Selective Reminding Test (FCSRT); Min score immediate recall trials=0; Max score immediate recall trials=48; Min score Delayed recall trials=0; Max score delayed recall trials=16. Higher scores on both trials mean a better outcome.

SECONDARY OUTCOMES:
Beck Depression Inventory II (BDI-II) (Depressive symptomatology) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the BDI-II; Min score=0; Max score=63; Higher scores mean a worse outcome.
World Health Organization Quality of Life - Bref (WHOQOL-Bref) (Quality of life) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the World Health Organization Quality of life-Bref (WHOQOL-Bref); Min score=0; Max score=100; Higher scores mean a better outcome.
Adults and Older Adults Functional Assessment Inventory (IAFAI) | Baseline (1 week before the beginning of the intervention), post-intervention (7 weeks) and follow-up (3-months)
  Change from baseline in the Adults and Older Adults Functional Assessment Inventory; (IAFAI). Min score=0; Max score=100; Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Casa de Saúde Câmara Pestana, Funchal, São Gonçalo, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camara J, Ferreira L, Faria AL, Vilar M, Bermudez I Badia S. Feasibility, Acceptability, and Preliminary Impact of Full-Body Interaction on Computerized Cognitive Training Based on Instrumental Activities of Daily Living: A Pilot Randomized Controlled Trial with Chronic Psychiatric Inpatients. Games Health J. 2022 Oct 11. doi: 10.1089/g4h.2021.0228. Online ahead of print. PMID 36251861

DOCUMENTS (1):
  • Study Protocol (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT05100849/Prot_000.pdf